CLINICAL TRIAL: NCT02390245
Title: Philadelphia Telemedicine Glaucoma Detection and Follow-Up Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wills Eye (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); Westat (Other); Public Health Management Corporation (Other); Philadelphia Department of Public Health (Other Government); Health Federation of Philadelphia (Other); Temple Physicians, Inc. (Industry)
Responsible Party: Principal Investigator, L. Jay Katz MD, MD, Wills Eye
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 14-441
Record Dates: First submitted 2015-03-11; First posted 2015-03-17 (Estimated); Results first posted 2022-03-11 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Glaucoma; Glaucoma Suspect; Diabetic Retinopathy; Ocular Hypertension; Cataract; Branch Retinal Vein Occlusion; Branch Retinal Arterial Occlusion; Central Retinal Vein Occlusion; Central Retinal Artery Occlusion; Epi-retinal Membrane; Macular Degeneration; Drusen; Loss of Vision
MeSH Terms: conditions — Glaucoma; Ocular Hypertension; Diabetic Retinopathy; Cataract; Retinal Vein Occlusion; Retinal Artery Occlusion; Macular Degeneration; Vision Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Phase 1: Telemedicine Screening Participants (Experimental): Participants across the Philadelphia, PA region were invited to participate in free eye screenings at primary care physician offices or health centers. Screenings included images of optic nerve and macula using non-contact, autofocus, hand-held fundus cameras (Volk Optical, Mentor, Ohio, USA) and measuring Intraocular Pressure (IOP) in millimeters of mercury (mm Hg) with non-contact rebound tonometers TA01I (ICare, Helsinki, Finland).
  Interventions: Other: Free Eye Screenings
- Phases 2 and 3: Enhanced Intervention Group (Experimental): From eye screening results (visit 1), Phase 2 includes participants requiring further evaluation received comprehensive eye exam to confirm diagnosis (visit 2). Following confirmation diagnosis, patients were randomized to the Enhanced Intervention Group and were referred to a general ophthalmologist for follow-up eye care. Patient navigation and a social worker and referred to a general ophthalmologist close to the current health center or primary care physician office where they received the non dilated eye exam. Prior to all follow-up visits, patients in the Enhanced Intervention Group were provided a scheduled appointment and received a personal phone call reminding them to attend. Patients received necessary interpretation services and educational materials.
  Phase 3. Includes following this group over a 5 year period for adherence to eye care.
  Interventions: Other: Enhanced Intervention
- Phases 2 and 3: Usual Care Group (Experimental): From eye screening results (visit 1), Phase 2 includes participants requiring further evaluation received comprehensive eye exam to confirm diagnosis (visit 2). Following confirmation diagnosis, patients were randomized to the Usual Care Group and were referred to a general ophthalmologist for follow-up eye care. These patients were scheduled for their initial follow-up visit based on the recommendations of our study physicians so the research team was able to track outcomes. This group represents a realistic choice currently available for patients. Practice patterns vary depending on the resources, staff time, and services available within each local ophthalmology practice.
  Phase 3. Includes following this group over a 5 year period for adherence to eye care.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Free Eye Screenings — This group will receive free eye screening and follow-up comprehensive ophthalmic exam if recommended.
  Arms: Phase 1: Telemedicine Screening Participants
Other: Enhanced Intervention — This group will receive ophthalmic referral and a navigator for assistance in scheduling appointments; confirming appointments via phone, mail, email and/or text message; arranging transportation through Customized Community Transportation (CCT) and Philadelphia Paratransit Service; and trained medical interpreters as needed.
  Arms: Phases 2 and 3: Enhanced Intervention Group
Other: Usual Care — This group will receive ophthalmic referral.
  Arms: Phases 2 and 3: Usual Care Group

SUMMARY:
The goal is to conduct a 5-year prospective, randomized controlled trial to test an innovative, community-based intervention using posterior and anterior fundus photography of the optic nerve and macula and intraocular eye pressure measurements to improve access and utilization of eye care to detect, treat, and manage high-risk patients with previously undiagnosed glaucoma and other eye diseases. Research shows that subject failure to attend follow-up eye care appointments diminishes any previous benefits of community screenings for glaucoma. Greater adherence to follow-up visits can reduce glaucomatous blindness.

DETAILED DESCRIPTION:
The project will be divided into following parts:

* Phase 1 will consist of recruiting patients from primary care offices and federally qualified health centers across Philadelphia and Chester counties. Using fundus photography of optic nerve and macula via telemedicine and measurement of intraocular pressure, eye disease will be detected at Visit 1, followed by a comprehensive eye exam by a glaucoma specialist in the primary care setting to confirm the diagnosis (Visit 2) of qualifying participants requiring further evaluation. Predictive accuracy of optic nerve images to detect glaucoma, glaucoma suspect and other eye diseases as confirmed by the comprehensive eye exam will be evaluated.
* Phase 2 will involve consenting, enrolling, and randomizing the qualifying participants confirmed by diagnosis at Visit 2 to either the Usual Care group or the Enhanced Intervention group and scheduling follow-up eye exams with a local, general ophthalmologist in an office-based setting (Visit 3). Enhanced intervention will use patient navigators and a social worker to reduce barriers to follow-up eye care.
* Phase 3 will involve monitoring the randomized participants attendance of proximal (1-2 months) and distal (3 years) follow-up care appointments (Visits 3-8) with a local ophthalmologist. Adherence to recommendations for follow-up eye care will be the primary outcome measure. A comprehensive estimation of intervention costs and cost-effectiveness of detecting eye diseases and vision impairment in a high-risk population will also be conducted. Protocols, materials, and results will be disseminated to other organizations, stakeholders and communities in order to expand detection of glaucoma, other eye diseases, and visual impairment, and to further refine these approaches.

ELIGIBILITY:
Inclusion Criteria:

* African-American, Hispanic, or Asian individuals over age 40
* Caucasian individuals over age 65
* Individuals of any ethnicity, over age 40 with a family history of glaucoma
* Individuals of any ethnicity, over age 40 with diabetes
* Individuals who meet one of the above criteria who have not seen an ophthalmologist in the past year

Exclusion Criteria:

Any patient with previously diagnosed glaucoma, glaucoma suspect, or eye diseases who is currently being followed by an ophthalmologist

-

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 906 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2020-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: L. J Katz, MD, Principal Investigator — Wills Eye Hospital; Lisa A Hark, PhD, Principal Investigator — Wills Eye Hospital; Julia A Haller, MD, Principal Investigator — Wills Eye Hospital
Locations (1):
- Wills Eye Glaucoma Service, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
A methods paper with year-1 baseline data and cost analysis has been published. Additional scientific manuscripts are under development.

REFERENCES:
- [Result] Hark LA, Katz LJ, Myers JS, Waisbourd M, Johnson D, Pizzi LT, Leiby BE, Fudemberg SJ, Mantravadi AV, Henderer JD, Zhan T, Molineaux J, Doyle V, Divers M, Burns C, Murchison AP, Reber S, Resende A, Bui TDV, Lee J, Crews JE, Saaddine JB, Lee PP, Pasquale LR, Haller JA. Philadelphia Telemedicine Glaucoma Detection and Follow-up Study: Methods and Screening Results. Am J Ophthalmol. 2017 Sep;181:114-124. doi: 10.1016/j.ajo.2017.06.024. Epub 2017 Jun 30. PMID 28673747
- [Result] Leiby BE, Hegarty SE, Zhan T, Myers JS, Katz LJ, Haller JA, Waisbourd M, Burns C, Divers M, Molineaux J, Henderer J, Brodowski C, Hark LA. A Randomized Trial to Improve Adherence to Follow-up Eye Examinations Among People With Glaucoma. Prev Chronic Dis. 2021 May 20;18:E52. doi: 10.5888/pcd18.200567. PMID 34014814
- [Derived] Hark LA, Myers JS, Ines A, Jiang A, Rahmatnejad K, Zhan T, Leiby BE, Hegarty S, Fudemberg SJ, Mantravadi AV, Waisbourd M, Henderer JD, Burns C, Divers M, Molineaux J, Pizzi LT, Murchison AP, Saaddine J, Pasquale LR, Haller JA, Katz LJ. Philadelphia Telemedicine Glaucoma Detection and Follow-up Study: confirmation between eye screening and comprehensive eye examination diagnoses. Br J Ophthalmol. 2019 Dec;103(12):1820-1826. doi: 10.1136/bjophthalmol-2018-313451. Epub 2019 Feb 15. PMID 30770354

RESULTS

PARTICIPANT FLOW:
Groups:
- Telemedicine Screening Participants - Phase 1: Phase I Participants recruited from diverse underserved locations across the Philadelphia region were invited for a free eye screening Visit 1 conducted at 14 locations by study team.
  Screenings consisted of noncontact, autofocus, hand-held fundus camera (Volk Optical, Mentor, Ohio, USA) to detect abnormalities on optic nerve and macula. Trained ocular technicians captured 2 posterior and 1 anterior images per eye (6 photographs).
  Intraocular pressure (IOP) in millimeters of mercury (mm Hg) was assessed with noncontact rebound tonometer TA01I (ICare, Helsinki, Finland). Single IOP taken for each eye. If IOP > 22 mm Hg, second IOP taken of that eye. If difference between 2 measurements < 2 mm Hg, average recorded. If difference between 2 measurements > 2 mm Hg, third measurement obtained, and median recorded.
  Visual acuity measured with correction, if patient had glasses or contact lenses, using digital acuity system ClearChart 2 (Reichert Technologies, Depew, New York, USA).
  Medical, family and ocular history recorded. Participants with suspicious findings, high eye pressure or unreadable images were invited back for complete eye examination Visit 2 at primary care physician offices to confirm diagnosis. If final IOP > 30 mm Hg, participant Fast Tracked to Visit 2.
- Enhanced Intervention Group - Phases 2/3: Phase II Included confirmation dilated eye exam (Visit 2) for qualifying participants with ocular hypertension or glaucoma. Participants were randomized into an Enhanced Intervention Group then referred to a general ophthalmologist for follow-up eye care. The Enhanced Intervention Group was assigned a patient navigator and social worker and scheduled for an initial follow-up visit based on recommendations from study physicians at Visit 2. Prior to all follow-up visits, participants were given a scheduled appointment and received personal phone call reminders. Patients received necessary interpretation services and educational materials.
  Phase III consisted of tracking the Enhanced Intervention Group for compliance of attending recommended ophthalmic visits after Visit 2 during a 5 year period. Tracking was performed by the research team.
- Usual Care Group - Phases 2/3: Phase II Included confirmation dilated eye exam (Visit 2) for qualifying participants with ocular hypertension or glaucoma. Participants were randomized into a Usual Care Group then referred to a general ophthalmologist for follow-up eye care. The Usual Care Group was scheduled for an initial follow-up visit based on recommendations from study physicians at Visit 2. This option represents a realistic choice currently available to patients. Practice patterns vary depending on resources, staff time, and services available within each local ophthalmology practice.
  Phase III consisted of tracking the Usual Care Group for compliance of attending recommended ophthalmic visits after Visit 2 during a 5 year period. Tracking was performed by the research team.
Period: Phase I. Telemedicine Screening
Arm/Group | Telemedicine Screening Participants - Phase 1 | Enhanced Intervention Group - Phases 2/3 | Usual Care Group - Phases 2/3
Started | 906 | 0 | 0
Completed | 906 | 0 | 0
Not Completed | 0 | 0 | 0
Period: Phase 2. Randomization Into 2 Groups
Arm/Group | Telemedicine Screening Participants - Phase 1 | Enhanced Intervention Group - Phases 2/3 | Usual Care Group - Phases 2/3
Started | 0 (Remaining 355 participants from Phase I Telemedicine Screening had normal eye examinations requiring no further follow-up.) | 275 | 276
Completed | 0 | 172 | 172
Not Completed | 0 | 103 | 104
Not completed — Lost to Follow-up | 0 | 103 | 104
Period: Phase 3. Ophthalmic Follow-up Adherence
Arm/Group | Telemedicine Screening Participants - Phase 1 | Enhanced Intervention Group - Phases 2/3 | Usual Care Group - Phases 2/3
Started | 0 | 172 | 172
Completed | 0 | 77 | 66
Not Completed | 0 | 95 | 106
Not completed — Lost to Follow-up | 0 | 95 | 106

BASELINE CHARACTERISTICS:
Population: Phase 1. Participants were recruited from diverse underserved locations across the Philadelphia region from community partners which included Public Health Management Corporation (4 centers), Philadelphia Department of Public Health (1 center), Health Federation of Philadelphia (2 centers), and Temple Physicians Inc (7 primary care offices). Offices and health centers were selected based on zip code. Qualifying participants were offered the option of Phase 2 and 3 participation.
Groups:
- Telemedicine Screening Participants - Phase 1: Phase 1: Participants from geographically underserved locations across the Philadelphia, PA region were invited to participate in a free glaucoma eye screening at their primary care physician offices or health centers which included taking images of optic nerve and macula using a non-contact, autofocus, hand-held fundus camera (Volk Optical, Mentor, Ohio, USA) and measuring Intraocular Pressure (IOP) in millimeters of mercury (mm Hg) with a non-contact rebound tonometer TA01I (ICare, Helsinki, Finland). Visual acuity was measured with correction, if patient had glasses or contact lenses, using the digital acuity system ClearChart 2 (Reichert Technologies, Depew, New York, USA) and medical, family and ocular history were recorded
Arm/Group | Telemedicine Screening Participants - Phase 1
Number analyzed (Participants) | 906
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 635
  >=65 years | 271
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 553
  Male | 353
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 123
  Not Hispanic or Latino | 770
  Unknown or Not Reported | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 49
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 550
  White | 154
  More than one race | 15
  Unknown or Not Reported | 137
Region of Enrollment [Number; unit: participants]
  United States | 906
Screening categories [Count of Participants; unit: Participants] — Participants were informed and invited ahead of scheduled screenings. During scheduled screenings, other individuals interested in participating were included as Walk-ins if inclusion/exclusion criteria was met.
  Participants
    Scheduled participants | 541
    Walk-in participants | 365

OUTCOME MEASURES:

1. Primary Outcome: Fundus Camera Images Via Telemedicine
Description: Phase I. Detection of glaucoma and other eye diseases using non contact, autofocus, hand-held fundus camera (Volk Optical, Mentor, Ohio, USA) with images of optic nerve and macula and confirmed at follow-up full dilated eye examination by ophthalmologists.
Time Frame: 1 hour eye exam
Measure: Count of Participants; unit: Participants
Groups:
- Telemedicine Screening Participants: Phase I. Participants recruited from diverse underserved locations across the Philadelphia region from community partners. Community partners included Public Health Management Corporation (4 centers), Philadelphia Department of Public Health (1 center), Health Federation of Philadelphia (2 centers), and Temple Physicians Inc (7 primary care offices). Offices and health centers selected based on zip code.
  Screenings consisted of a non contact, autofocus, hand-held fundus camera (Volk Optical, Mentor, Ohio, USA) to center images on the optic nerve and macula. Trained ocular technicians captured 2 posterior and 1 anterior images per eye (6 total photographs).
  Intraocular pressure (IOP) in millimeters of mercury (mm Hg) was assessed with non contact rebound tonometer TA01I (ICare, Helsinki, Finland). Single IOP taken for each eye. If IOP > 22 mm Hg, a second IOP was taken of that eye. If difference between 2 measurements < 2 mm Hg, average was recorded. If difference between 2 measurements > 2 mm Hg, a third measurement was obtained, and median was recorded. If final IOP > 30 mm Hg, participant was Fast Tracked to Visit 2.
  Visual acuity measured with correction, if patient had glasses or contact lenses, using the digital acuity system ClearChart 2 (Reichert Technologies, Depew, New York, USA).
  Medical, family and ocular history were recorded.
Arm/Group | Telemedicine Screening Participants
Number analyzed (Participants) | 906
Participants
  Normal fundus images | 355
  Abnormal fundus images | 384
  Unreadable images | 167

2. Primary Outcome: Intraocular Pressure
Description: Phase I. Intraocular pressure (IOP) as measured in millimeters of mercury (mm Hg) with non contact rebound tonometer TA01I (ICare, Helsinki, Finland). Single IOP taken for each eye. If IOP > 22 mm Hg, a second IOP was taken of that eye. If difference between 2 measurements < 2 mm Hg, average was recorded. If difference between 2 measurements > 2 mm Hg, a third measurement was obtained, and median was recorded. If final IOP > 30 mm Hg, participant was Fast Tracked to Visit 2.
Time Frame: 1 hour eye exam
Measure: Count of Participants; unit: Participants
Arm/Group | Telemedicine Screening Participants
Number analyzed (Participants) | 906
Participants
  IOP 30-34 mmHg | 10
  IOP 35-39 mmHg | 3
  IOP >39 mmHg | 2
  IOP 22-29 mmHg | 728
  IOP <21 mmHg | 163

3. Primary Outcome: Diagnostic Image Confirmation by Ophthalmologist
Description: Phase I. Confirmation of telemedicine screen Visit 1 findings with a diagnosis following complete dilated eye examination and visual field by study team and Ophthalmologist at Visit 2.
Time Frame: 1 hour eye examination
Population: 355 of 906 participants of telemedicine screen Visit 1 did not require follow-up visits.
Measure: Count of Participants; unit: Participants
Groups:
- Telemedicine Screening Participants: Phase I. Participants with suspicious findings, high eye pressure or unreadable images from the telemedicine screening Visit 1 were referred for a complete dilated eye examination and visual field by study team and Ophthalmologist at Visit 2 within 6 months.
Arm/Group | Telemedicine Screening Participants
Number analyzed (Participants) | 551
Participants
  Glaucoma | 38
  Glaucoma Suspects | 159
  Ocular Hypertension | 25
  Anatomically narrow angles | 23
  IOP >30 mmHg | 15
  Other retinal diseases | 84
  Declined or Lost to Follow-up | 207

4. Secondary Outcome: Adherence to Follow-up Ophthalmic Care.
Description: Phase III: Compliance by participants was monitored for attending recommended follow-up eye care with ophthalmologist/optometrist in the Usual Care and Intervention Groups during a 5 year period. Follow-up visit recommendations were not predetermined, they were at the ophthalmologist/optometrist discretion and /or according to clinical practice. Adherence was achieved when completing visit 3 within 12 months of randomization. Visit 4 adherence was achieved if recommended follow-up of 3-4 months, 6 months or 12 months were completed within 6, 12 or 15 months, respectively.
Time Frame: 5 year follow-up period.
Measure: Count of Participants; unit: Participants
Groups:
- Enhanced Intervention Group - Phase III: Phase III consisted of tracking the Enhanced Intervention Group for compliance of attending recommended ophthalmic visits after Visit 2 during a 5 year period. The Enhanced Intervention Group was assigned a patient navigator and social worker throughout study period. Prior to all follow-up visits, participants were given a scheduled appointment and received personal phone call reminders. Patients received necessary interpretation services and educational materials.
  Tracking was performed by the research team.
- Usual Care Group - Phase III: Phase III consisted of tracking the Usual Care Group for compliance of attending recommended ophthalmic visits after Visit 2 during a 5 year period. Tracking was performed by the research team.
Arm/Group | Enhanced Intervention Group - Phase III | Usual Care Group - Phase III
Number analyzed (Participants) | 172 | 172
Participants
  Attended Visit 3 within 12 months of randomization | 128 | 67
  Attended visits in Year 1 according to ophthalmologist/optometrist recommendation | 32 | 14
  Attended Visit 4 according to ophthalmologist/optometrist recommendation | 97 | 39
  Adherence to follow-up visits in Year 2 according to ophthalmologist/optometrist recommendation | 27 | 9
  Adherence to follow-up visits in Year 3 according to ophthalmologist/optometrist recommendation | 5 | 1

ADVERSE EVENTS:
Time Frame: Phases 1 and 2: 1 hour eye examinations. Phase 3: 5 year follow-up period.
Description: Of the 551 Phase 1 participants qualifying for Phase 2 (Visit 2), 209 were Lost to Follow-up.
Groups:
- Phase 1: Telemedicine Screening Participants: Phase 1. 906 participants completed telemedicine screening with non contact fundus images, non contact intraocular pressure measurements, visual acuity and history recorded.
- Phases 2/3: Enhanced Intervention Group: Phase 2. 172 participants completing Visit 2 then randomized to the Enhanced Intervention Group for follow-up eye care.
  Phase 3. Includes following this group over a 5 year period for adherence to eye care.
- Phases 2/3: Usual Care Group: Phase 2. 172 participants completing Visit 2 then randomized to the Usual Care Group for follow-up eye care.
  Phase 3. Includes following this group over a 5 year period for adherence to eye care.
Arm/Group | Phase 1: Telemedicine Screening Participants | Phases 2/3: Enhanced Intervention Group | Phases 2/3: Usual Care Group
All-Cause Mortality (participants affected / at risk) | 0/906 | 0/172 | 0/172
Serious Adverse Events (participants affected / at risk) | 0/906 | 0/172 | 0/172
Other Adverse Events (participants affected / at risk) | 0/906 | 0/172 | 0/172

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-22): https://cdn.clinicaltrials.gov/large-docs/45/NCT02390245/Prot_SAP_000.pdf